CLINICAL TRIAL: NCT05366010
Title: Evaluation of Oscillation and Lung Expansion (OLE) Using The Volara® System for Treatment of Respiratory Complications in Patients With Neuromuscular Disease in the Home Setting
Brief Title: Oscillation and Lung Expansion (OLE) Therapy for Treatment of Neuromuscular Disease (NMD) Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Baxter Healthcare Corporation (Industry)
Collaborators: Science 37 (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-RR-2020-005
Record Dates: First submitted 2022-04-27; First posted 2022-05-09 (Actual); Results first posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Neuromuscular Diseases
MeSH Terms: conditions — Neuromuscular Diseases | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Study subjects will serve as their own control. Medical records will be reviewed for each study subject for the twelve-month period prior to initiation of OLE therapy. The study will compare the frequency of exacerbations experienced prior to treatment with OLE to the frequency of exacerbations experienced in the active treatment period, during which study subjects receive treatment with The Volara® System. In addition, specific healthcare utilization indicators including hospitalizations, antibiotic use, and emergency department (ED) visits for pulmonary complications will be documented for each study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Intervention (Experimental): Intervention time period, during which all subjects receive OLE therapy as their airway clearance intervention
  Interventions: Device: Oscillation and Lung Expansion (OLE) therapy

INTERVENTIONS:
Device: Oscillation and Lung Expansion (OLE) therapy — Respiratory airway clearance intervention including continuous high-frequency oscillation and continuous positive expiratory pressure

SUMMARY:
The study will be a non-randomized open label pilot study comparing a retrospective control period to an active treatment period with oscillation and lung expansion (OLE) therapy.

DETAILED DESCRIPTION:
The study is a decentralized trial. All data will be collected in the patients' homes. The primary objective of the study is to evaluate the impact of OLE to treat respiratory complications of neuromuscular disease patients. The frequency of pulmonary exacerbations and other clinical outcome measures will be assessed to determine the effect of consistent OLE therapy.

ELIGIBILITY:
Patients who met all the following inclusion criteria are included in the study:

* Documented diagnosis of neuromuscular disease (NMD) or neurological disorder.
* Age 5 to 80 years.
* History of one or more respiratory exacerbations in the past 6 months or two or more respiratory exacerbations in the past 12 months, which required unplanned or unscheduled medical intervention.
* Ability to perform Oscillation and Lung Expansion (OLE) therapy as directed.
* Signed informed consent (and assent if minor patient).

Patients who meet any of the following criteria will be excluded from the study:

* Diagnosis with rapidly progressing NMD such as certain types of Motor Neuron Disease (MND).
* Requirement for continuous mechanical ventilation.
* Anticipated requirement for respiratory related hospitalization within the next six months.
* History of pneumothorax within the past 6 months.
* History of hemoptysis requiring embolization within past 12 months.
* Pregnancy.
* Home use of OLE therapy within the past 12 months.
* Inability or unwillingness to perform OLE therapy or study procedures as required.

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-02-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Science 37, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Retrospective data was collected from a total of 41 patients. Two patients died prior to study start. Thus, these two patients were excluded from any safety analyses as they had no exposure to the Volara System.
Period: Overall Study
Arm/Group | Intervention
Started | 39
Completed | 33
Not Completed | 6
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 1
Not completed — Lost to Follow-up | 2
Not completed — Screen Failure | 2

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.4 (15.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 5
  White | 19
  More than one race | 2
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Exacerbations of Pulmonary Disease Requiring Medical Intervention
Description: Exacerbation of pulmonary disease is a worsening of pulmonary condition or an event requiring one or more of the following:
  * Hospitalization
  * Emergency Department visit
  * Unscheduled antibiotics
  * Unscheduled outpatient visit
Time Frame: 6 months pre-treatment and 6 months post-treatment with the Volara System
Measure: Mean (Standard Deviation); unit: Exacerbations
Arm/Group | Intervention
Number analyzed (Participants) | 33
Exacerbations
  6 months pre-treatment | 1.0 (0.81)
  Volara active treatment | 1.2 (1.39)

2. Secondary Outcome: Slow Vital Capacity
Description: Slow Vital Capacity is the maximum volume that the subject can exhale in a single breath, following full inspiration. The measure is taken using a slow consistent exhalation.
Time Frame: Baseline and monthly for 6 months
Population: Pulmonary Function Tests were analyzed for the Full Analysis Set (N=33). Of the Full Analysis Set, 12 subjects had data available for Slow Vital Capacity. The number of participants analyzed at each timepoint reflects the patients who were strong enough and had coordination to have this measurement taken.
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | Intervention
Number analyzed (Participants) | 12
Litres
  Baseline: number analyzed (Participants) | 10
  Baseline | 1.523 (0.7664)
  1 month: number analyzed (Participants) | 8
  1 month | 1.609 (0.6891)
  2 months: number analyzed (Participants) | 7
  2 months | 1.693 (0.6684)
  3 months: number analyzed (Participants) | 9
  3 months | 1.741 (0.6763)
  4 months: number analyzed (Participants) | 7
  4 months | 1.407 (0.6580)
  5 months: number analyzed (Participants) | 6
  5 months | 1.498 (0.5858)
  6 months: number analyzed (Participants) | 7
  6 months | 1.601 (0.4604)

3. Secondary Outcome: Peak Cough Flow
Description: Peak Cough Flow is a pulmonary function measure that evaluates maximum peak flow generated during a cough maneuver. It will be measured with a hand-held spirometer.
Time Frame: Baseline and monthly for 6 months
Population: Pulmonary Function Tests were analyzed for the Full Analysis Set (N=33). Of the Full Analysis Set, 10 subjects had data available for Peak Cough Flow. The number of participants analyzed at each timepoint reflects the patients who were strong enough and had coordination to have this measurement taken.
Measure: Mean (Standard Deviation); unit: Litres per second
Arm/Group | Intervention
Number analyzed (Participants) | 10
Litres per second
  Baseline: number analyzed (Participants) | 7
  Baseline | 2.121 (1.4399)
  1 month: number analyzed (Participants) | 6
  1 month | 2.730 (1.3391)
  2 months: number analyzed (Participants) | 2
  2 months | 2.595 (0.0778)
  3 months: number analyzed (Participants) | 5
  3 months | 2.874 (0.6911)
  4 months: number analyzed (Participants) | 3
  4 months | 3.297 (0.5543)
  5 months: number analyzed (Participants) | 3
  5 months | 3.327 (0.9673)
  6 months: number analyzed (Participants) | 3
  6 months | 2.153 (1.6887)

4. Secondary Outcome: Resting Oxygen Saturation
Description: Oxygen Saturation will be measured while the subject is resting using a hand-held oximeter.
Time Frame: Baseline and monthly for 6 months
Population: Pulmonary Function Tests were analyzed for the Full Analysis Set (N=33). Of the Full Analysis Set, 22 subjects had data available for Resting Oxygen Saturation. The number of participants analyzed at each timepoint reflects the patients who were strong enough and had coordination to have this measurement taken.
Measure: Mean (Standard Deviation); unit: percentage oxygen saturation
Arm/Group | Intervention
Number analyzed (Participants) | 22
percentage oxygen saturation
  Baseline: number analyzed (Participants) | 11
  Baseline | 95.68 (1.978)
  1 month: number analyzed (Participants) | 9
  1 month | 96.78 (1.986)
  2 months: number analyzed (Participants) | 7
  2 months | 96.57 (2.699)
  3 months: number analyzed (Participants) | 11
  3 months | 96.73 (1.794)
  4 months: number analyzed (Participants) | 9
  4 months | 96.11 (2.759)
  5 months: number analyzed (Participants) | 6
  5 months | 97.00 (2.000)
  6 months: number analyzed (Participants) | 11
  6 months | 95.64 (3.641)

5. Secondary Outcome: Maximal Inspiratory Pressure
Description: Maximal Inspiratory Pressure is the maximum force (measured in centimeters of water [cmH2O]) that the subject can generate during an inspiratory effort.
Time Frame: Baseline and monthly for 6 months
Population: Pulmonary Function Tests were analyzed for the Full Analysis Set (N=33). Of the Full Analysis Set, 11 subjects had data available for Maximal Inspiratory Pressure. The number of participants analyzed at each timepoint reflects the patients who were strong enough and had coordination to have this measurement taken.
Measure: Mean (Standard Deviation); unit: centimeters of water
Arm/Group | Intervention
Number analyzed (Participants) | 11
centimeters of water
  Baseline: number analyzed (Participants) | 10
  Baseline | -40.7 (16.56)
  1 month: number analyzed (Participants) | 7
  1 month | -45.7 (16.18)
  2 months: number analyzed (Participants) | 7
  2 months | -46.3 (17.86)
  3 months: number analyzed (Participants) | 8
  3 months | -48.6 (16.81)
  4 months: number analyzed (Participants) | 6
  4 months | -42.3 (18.29)
  5 months: number analyzed (Participants) | 6
  5 months | -42.8 (21.91)
  6 months: number analyzed (Participants) | 6
  6 months | -50.8 (12.81)

6. Secondary Outcome: Number of Hospital Admissions
Description: Number of hospital admissions for respiratory complications.
Time Frame: 6 months pre-treatment with the Volara System and 6 months post-treatment with the Volara System
Measure: Mean (Standard Deviation); unit: number of visits
Arm/Group | Intervention
Number analyzed (Participants) | 33
number of visits
  6 months pre-treatment | 0.5 (0.67)
  Volara active treatment | 0.4 (0.75)

7. Secondary Outcome: Total Hospital Length of Stay
Description: Number of inpatient hospital days for respiratory complications
Time Frame: 6 months pre-treatment with the Volara System and 6 months post-treatment with the Volara System
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention
Number analyzed (Participants) | 33
days
  6 months pre-treatment | 5.2 (7.90)
  Volara active treatment | 1.7 (3.19)

8. Secondary Outcome: Number of Intensive Care Unit (ICU) Admissions
Description: Number of ICU admissions for respiratory complications.
Time Frame: 6 months pre-treatment with the Volara System and 6 months post-treatment with the Volara System
Measure: Mean (Standard Deviation); unit: Number of visits
Arm/Group | Intervention
Number analyzed (Participants) | 33
Number of visits
  6 months pre-treatment | 0.2 (0.55)
  Volara active treatment | 0.2 (0.53)

9. Secondary Outcome: Total Intensive Care Unit (ICU) Length of Stay
Description: Number of ICU hospital days for respiratory complications
Time Frame: 6 months pre-treatment with the Volara System and 6 months post-treatment with the Volara System
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention
Number analyzed (Participants) | 33
days
  6 months pre-treatment | 1.9 (5.42)
  Volara active treatment | 0.8 (2.41)

10. Secondary Outcome: Number of Outpatient Visits for Pulmonary Complications
Description: Number of unscheduled Physician's office visits, urgent care visits, and emergency department (ED) visits.
Time Frame: 6 months pre-treatment and 6 months post-treatment with the Volara System
Measure: Mean (Standard Deviation); unit: Number of visits
Arm/Group | Intervention
Number analyzed (Participants) | 33
Number of visits
  6 months pre-treatment | 0.7 (0.82)
  Volara active treatment | 0.9 (1.20)

11. Secondary Outcome: Total Number of Antibiotic Use Days During Episodes for Respiratory Infection
Description: The total number of antibiotic use days includes any of the following: intravenous (IV) antibiotic days, oral antibiotic days, and nebulized antibiotic days.
Time Frame: 6 months pre-treatment and 6 months post-treatment with the Volara System
Measure: Mean (Standard Deviation); unit: Number of days
Arm/Group | Intervention
Number analyzed (Participants) | 33
Number of days
  6 months pre-treatment | 6.6 (8.04)
  Volara active treatment | 4.5 (7.57)

12. Secondary Outcome: Adherence to Treatment Regimen: Average Daily Volara System Usage
Description: Adherence to the OLE treatment regimen was presented as Average Daily Volara System Usage. This was calculated by dividing the total minutes of device use by the total number of days the subject had the device.
Time Frame: Total number of days the subject had the device (approximately up to 6 months of OLE therapy)
Population: Device usage information was only available for 18 of the 33 subjects as the remaining subjects did not return the Volara System. Some subjects retained the device beyond the 6-month active treatment period.
Measure: Mean (Standard Deviation); unit: minutes/day
Arm/Group | Intervention
Number analyzed (Participants) | 18
minutes/day | 15.1 (13.7)

13. Secondary Outcome: Impact of OLE Therapy on Patient Quality of Life Using the Respiratory Complaints Domain of the Severe Respiratory Insufficiency (SRI) Questionnaire
Description: Severe Respiratory Insufficiency (SRI) questionnaire administered at baseline, and at 1, 3 and 6 months. The total score can range from a minimum of 0 to a maximum of 100 with higher values indicating a better health-related quality of life according to content of the scale.
Time Frame: Baseline, and after 1 month, 3 months, and 6 months of therapy using the Volara System
Population: All responses obtained are presented. Some patients did not provide feedback at certain follow-up visits.
Measure: Mean (Standard Deviation); unit: Score on SRI scale
Arm/Group | Intervention
Number analyzed (Participants) | 33
Score on SRI scale
  Baseline: number analyzed (Participants) | 31
  Baseline | 45.654 (22.6888)
  1 month: number analyzed (Participants) | 29
  1 month | 57.000 (21.0432)
  3 months: number analyzed (Participants) | 28
  3 months | 59.953 (22.4735)
  6 months: number analyzed (Participants) | 27
  6 months | 63.390 (21.2530)

14. Secondary Outcome: Satisfaction With Current Airway Clearance Therapy at Baseline
Description: Satisfaction is assessed through a questionnaire administered at baseline. Seven satisfaction questions are assessed using a Five-point Likert Scale. Total score is from 5 to 35, with 35 indicating the highest satisfaction.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Groups:
- Intervention: Intervention time period, during which subjects received their current airway clearance intervention.
Arm/Group | Intervention
Number analyzed (Participants) | 33
Participants
  Q1R1. It is so difficult to use the current airway clearance therapy that I do not want to use it | 0
  Q1R2. It is very difficult to use the current airway clearance therapy | 0
  Q1R3. It is moderately difficult to use the current airway clearance therapy | 7
  Q1R4. It is fairly easy to use the current airway clearance therapy | 14
  Q1R5. It is very easy to use the current airway clearance therapy | 5
  Q1R0. No answer on ease/difficulty of using the current airway clearance therapy | 7
  Q2R1. It is so difficult to tolerate the current airway clearance therapy that I don't want to do it | 0
  Q2R2. It is very difficult to tolerate the current airway clearance therapy | 1
  Q2R3. It is moderately difficult to tolerate the current airway clearance therapy | 6
  Q2R4. It is fairly easy to tolerate the current airway clearance therapy | 12
  Q2R5. It is very easy to tolerate the current airway clearance therapy | 6
  Q2R0. No answer on ease/difficulty of tolerating the current airway clearance therapy | 8
  Q3R1. I never miss therapy with the current airway clearance therapy | 12
  Q3R2. I miss therapy once a week | 7
  Q3R3. I miss therapy twice a week | 2
  Q3R4. I miss therapy three times a week | 3
  Q3R5. I miss therapy four or more times a week | 1
  Q3R0. No response on frequency of missing therapy per week | 8
  Q4R1. The current airway clearance is not effective as I never bring up sputum with therapy | 2
  Q4R2. The current airway clearance therapy is effective sometimes | 11
  Q4R3. The current airway clearance therapy is mostly effective | 6
  Q4R4. The current airway clearance therapy is almost always effective | 5
  Q4R5. I always bring up sputum with therapy | 2
  Q4R0. No answer on effectiveness of current airway clearance therapy on bringing up sputum | 7
  Q5R1. I always feel short of breath | 0
  Q5R2. I frequently have shortness of breath episodes | 2
  Q5R3. I have some shortness of breath episodes | 5
  Q5R4. I have a few shortness of breath episodes | 15
  Q5R5. I never have shortness of breath | 3
  Q5R0. No answer on effect of current airway clearance therapy on breathing | 8
  Q6R1. I do not feel the current airway clearance therapy helps my lungs stay healthy | 1
  Q6R2. I am unsure if this therapy helps my lungs stay healthy | 0
  Q6R3. This therapy seems somewhat helpful helpful for my lungs | 10
  Q6R4. I feel this therapy helps my lungs stay healthy | 10
  Q6R5. I definitely feel this therapy helps my lungs stay healthy | 4
  Q6R0. No answer on whether patients feel the current therapy helps their lungs feel healthy | 8
  Q7R1. My ability to perform daily tasks has definitely not improved | 1
  Q7R2. My ability to perform daily tasks has not improved | 2
  Q7R3. I am unsure if my ability to perform daily tasks has improved | 8
  Q7R4. I have had some improvement in ability to perform daily tasks | 13
  Q7R5. I have had significant improvement in ability to perform daily tasks | 1
  Q7R0. No answer on effect of current therapy on ability to perform daily tasks | 8

15. Secondary Outcome: Satisfaction With OLE Therapy After 1 Month of Using the Volara System
Description: Satisfaction is assessed through a questionnaire administered after 1 month of therapy using the Volara System. Eight satisfaction questions are assessed using a Five-point Likert Scale. Total score is from 5 to 40, with 40 indicating the highest satisfaction.
Time Frame: After 1 month of using the Volara System
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 33
Participants
  Q1R1. It is so difficult to use the Volara System that I do not want to use it | 0
  Q1R2. It is very difficult to use the Volara System | 1
  Q1R3. It is moderately difficult to use the Volara System | 0
  Q1R4. It is fairly easy to use the Volara System | 15
  Q1R5. It is very easy to use the Volara System | 15
  Q1R0. No answer on ease/difficulty of using the Volara System | 2
  Q2R1. It is so difficult to tolerate therapy with the Volara System that I don't want to do it | 0
  Q2R2. It is very difficult to tolerate therapy with the Volara System | 2
  Q2R3. It is moderately difficult to tolerate therapy with the Volara System | 3
  Q2R4. It is fairly easy to tolerate therapy with the Volara System | 17
  Q2R5. It is very easy to tolerate therapy with the Volara System | 9
  Q2R0. No answer on ease/difficulty of tolerating therapy with the Volara System | 2
  Q3R1. I never miss therapy | 17
  Q3R2. I miss therapy once a week | 8
  Q3R3. I miss therapy twice a week | 1
  Q3R4. I miss therapy three times a week | 4
  Q3R5. I miss therapy four or more times a week | 0
  Q3R0. No response on frequency of missing therapy per week | 3
  Q4R1. The therapy is not effective as I never bring up sputum with therapy | 3
  Q4R2. The therapy is effective sometimes | 8
  Q4R3. The therapy is mostly effective | 11
  Q4R4. The therapy is almost always effective | 6
  Q4R5. I always bring up sputum with therapy | 3
  Q4R0. No answer on effectiveness of therapy in bringing up sputum | 2
  Q5R1. I always feel short of breath | 0
  Q5R2. I frequently have shortness of breath episodes | 0
  Q5R3. I have some shortness of breath episodes | 7
  Q5R4. I have a few shortness of breath episodes | 19
  Q5R5. I never have shortness of breath | 5
  Q5R0. No answer on effect of therapy on breathing | 2
  Q6R1. I do not feel the therapy helps my lungs stay healthy | 0
  Q6R2. I am unsure if this therapy helps my lungs stay healthy | 3
  Q6R3. This therapy seems somewhat helpful helpful for my lungs | 7
  Q6R4. I feel this therapy helps my lungs stay healthy | 15
  Q6R5. I definitely feel this therapy helps my lungs stay healthy | 5
  Q6R0. No answer on whether patients feel the therapy helps their lungs feel healthy | 3
  Q7R1. My ability to perform daily tasks has definitely not improved | 0
  Q7R2. My ability to perform daily tasks has not improved | 3
  Q7R3. I am unsure if my ability to perform daily tasks has improved | 14
  Q7R4. I have had some improvement in ability to perform daily tasks | 10
  Q7R5. I have had significant improvement in ability to perform daily tasks | 2
  Q7R0. No answer on effect of current therapy on ability to perform daily tasks | 4
  Q8R1. I do not want to continue. I strongly prefer to use my previous therapy | 0
  Q8R2. I prefer to use my previous therapy | 2
  Q8R3. I do not have a preference on which therapy I use | 3
  Q8R4. I prefer to continue to do therapy with the Volara System | 17
  Q8R5. I strongly prefer to continue to do therapy with the Volara System | 9
  Q8R0. No answer given on therapy preference | 2

16. Secondary Outcome: Satisfaction With OLE Therapy After 3 Months of Using the Volara System
Description: Satisfaction is assessed through a questionnaire administered after 3 months of therapy using the Volara System. Eight satisfaction questions are assessed using a Five-point Likert Scale. Total score is from 5 to 40, with 40 indicating the highest satisfaction.
Time Frame: After 3 months of using the Volara System
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 33
Participants
  Q1R1. It is so difficult to use the Volara System that I do not want to use it | 0
  Q1R2. It is very difficult to use the Volara System | 0
  Q1R3. It is moderately difficult to use the Volara System | 1
  Q1R4. It is fairly easy to use the Volara System | 15
  Q1R5. It is very easy to use the Volara System | 13
  Q1R0. No answer on ease/difficulty of using the Volara System | 4
  Q2R1. It is so difficult to tolerate therapy with the Volara System that I don't want to do it | 0
  Q2R2. It is very difficult to tolerate therapy with the Volara System | 0
  Q2R3. It is moderately difficult to tolerate therapy with the Volara System | 4
  Q2R4. It is fairly easy to tolerate therapy with the Volara System | 15
  Q2R5. It is very easy to tolerate therapy with the Volara System | 10
  Q2R0. No answer on ease/difficulty of tolerating therapy with the Volara System | 4
  Q3R1. I never miss therapy | 14
  Q3R2. I miss therapy once a week | 12
  Q3R3. I miss therapy twice a week | 2
  Q3R4. I miss therapy three times a week | 1
  Q3R5. I miss therapy four or more times a week | 0
  Q3R0. No response on frequency of missing therapy per week | 4
  Q4R1. The therapy is not effective as I never bring up sputum with therapy | 2
  Q4R2. The therapy is effective sometimes | 9
  Q4R3. The therapy is mostly effective | 5
  Q4R4. The therapy is almost always effective | 9
  Q4R5. I always bring up sputum with therapy | 4
  Q4R0. No answer on effectiveness of therapy in bringing up sputum | 4
  Q5R1. I always feel short of breath | 0
  Q5R2. I frequently have shortness of breath episodes | 1
  Q5R3. I have some shortness of breath episodes | 3
  Q5R4. I have a few shortness of breath episodes | 14
  Q5R5. I never have shortness of breath | 10
  Q5R0. No answer on effect of therapy on breathing | 5
  Q6R1. I do not feel the therapy helps my lungs stay healthy | 1
  Q6R2. I am unsure if this therapy helps my lungs stay healthy | 2
  Q6R3. This therapy seems somewhat helpful helpful for my lungs | 7
  Q6R4. I feel this therapy helps my lungs stay healthy | 12
  Q6R5. I definitely feel this therapy helps my lungs stay healthy | 7
  Q6R0. No answer on whether patients feel the therapy helps their lungs feel healthy | 4
  Q7R1. My ability to perform daily tasks has definitely not improved | 0
  Q7R2. My ability to perform daily tasks has not improved | 1
  Q7R3. I am unsure if my ability to perform daily tasks has improved | 12
  Q7R4. I have had some improvement in ability to perform daily tasks | 11
  Q7R5. I have had significant improvement in ability to perform daily tasks | 1
  Q7R0. No answer on effect of current therapy on ability to perform daily tasks | 8
  Q8R1. I do not want to continue. I strongly prefer to use my previous therapy | 1
  Q8R2. I prefer to use my previous therapy | 1
  Q8R3. I do not have a preference on which therapy I use | 5
  Q8R4. I prefer to continue to do therapy with the Volara System | 14
  Q8R5. I strongly prefer to continue to do therapy with the Volara System | 8
  Q8R0. No answer given on therapy preference | 4

17. Secondary Outcome: Satisfaction With OLE Therapy After 6 Months of Using the Volara System
Description: Satisfaction is assessed through a questionnaire administered after 6 months of therapy using the Volara System. Eight satisfaction questions are assessed using a Five-point Likert Scale. Total score is from 5 to 40, with 40 indicating the highest satisfaction.
Time Frame: After 6 months of using the Volara System
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 33
Participants
  Q1R1. It is so difficult to use the Volara System that I do not want to use it | 0
  Q1R2. It is very difficult to use the Volara System | 2
  Q1R3. It is moderately difficult to use the Volara System | 1
  Q1R4. It is fairly easy to use the Volara System | 13
  Q1R5. It is very easy to use the Volara System | 11
  Q1R0. No answer on ease/difficulty of using the Volara System | 6
  Q2R1. It is so difficult to tolerate therapy with the Volara System that I don't want to do it | 1
  Q2R2. It is very difficult to tolerate therapy with the Volara System | 2
  Q2R3. It is moderately difficult to tolerate therapy with the Volara System | 3
  Q2R4. It is fairly easy to tolerate therapy with the Volara System | 14
  Q2R5. It is very easy to tolerate therapy with the Volara System | 7
  Q2R0. No answer on ease/difficulty of tolerating therapy with the Volara System | 6
  Q3R1. I never miss therapy | 13
  Q3R2. I miss therapy once a week | 7
  Q3R3. I miss therapy twice a week | 2
  Q3R4. I miss therapy three times a week | 4
  Q3R5. I miss therapy four or more times a week | 1
  Q3R0. No response on frequency of missing therapy per week | 6
  Q4R1. The therapy is not effective as I never bring up sputum with therapy | 2
  Q4R2. The therapy is effective sometimes | 11
  Q4R3. The therapy is mostly effective | 7
  Q4R4. The therapy is almost always effective | 4
  Q4R5. I always bring up sputum with therapy | 3
  Q4R0. No answer on effectiveness of therapy in bringing up sputum | 6
  Q5R1. I always feel short of breath | 0
  Q5R2. I frequently have shortness of breath episodes | 2
  Q5R3. I have some shortness of breath episodes | 3
  Q5R4. I have a few shortness of breath episodes | 12
  Q5R5. I never have shortness of breath | 8
  Q5R0. No answer on effect of therapy on breathing | 8
  Q6R1. I do not feel the therapy helps my lungs stay healthy | 1
  Q6R2. I am unsure if this therapy helps my lungs stay healthy | 2
  Q6R3. This therapy seems somewhat helpful helpful for my lungs | 3
  Q6R4. I feel this therapy helps my lungs stay healthy | 13
  Q6R5. I definitely feel this therapy helps my lungs stay healthy | 8
  Q6R0. No answer on whether patients feel the therapy helps their lungs feel healthy | 6
  Q7R1. My ability to perform daily tasks has definitely not improved | 2
  Q7R2. My ability to perform daily tasks has not improved | 4
  Q7R3. I am unsure if my ability to perform daily tasks has improved | 7
  Q7R4. I have had some improvement in ability to perform daily tasks | 7
  Q7R5. I have had significant improvement in ability to perform daily tasks | 5
  Q7R0. No answer on effect of current therapy on ability to perform daily tasks | 8
  Q8R1. I do not want to continue. I strongly prefer to use my previous therapy | 3
  Q8R2. I prefer to use my previous therapy | 2
  Q8R3. I do not have a preference on which therapy I use | 2
  Q8R4. I prefer to continue to do therapy with the Volara System | 9
  Q8R5. I strongly prefer to continue to do therapy with the Volara System | 8
  Q8R0. No answer given on therapy preference | 9

ADVERSE EVENTS:
Time Frame: Duration of participation for enrolled patients ranged from 16 days to 354 days.
Description: All-Cause Mortality was assessed in all enrolled patients. Adverse events were assessed for the patients who received treatment using the Volara System.
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 2/41
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 2/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=33)
Seizure (Nervous system disorders) | 1 (1)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
It may be that only the first pulmonary exacerbation in the 6 months before using Volara was recorded for patient enrollment.

Early termination led to a small number of patients being analyzed. Some patients were unable to undergo all planned analyses, such as Pulmonary Function Tests.

Selected patient population was broad in age and disease implying variability in disease trajectory and/or severity at enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor reserves the right of prior review and approval of data from this study relative to the potential release of proprietary information to any publication or for any presentation.

DOCUMENTS (2):
  • Study Protocol (2022-05-11): https://cdn.clinicaltrials.gov/large-docs/10/NCT05366010/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-28): https://cdn.clinicaltrials.gov/large-docs/10/NCT05366010/SAP_001.pdf